CLINICAL TRIAL: NCT04292782
Title: Caudal Epidural Block Compared to Anterior Quadratus Lumborum Block for Pediatric Hip Surgery
Brief Title: Quadratus Lumborum Block for Pediatric Hip Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Tunis El Manar (Other)
Collaborators: Institut Kassab d'Orthopédie (Other)
Responsible Party: Principal Investigator, Olfa kaabachi, MD, Professor, University Tunis El Manar
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CE-IMKO 104/2019
Record Dates: First submitted 2020-02-23; First posted 2020-03-03 (Actual); Last update posted 2024-02-13 (Actual); Status verified 2024-02

CONDITIONS: Hip Dislocation, Congenital; Postoperative Pain; Anesthesia
Keywords: hip dislocation; regional anesthesia; surgery
MeSH Terms: conditions — Hip Dislocation, Congenital; Pain, Postoperative; Hip Dislocation

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CAUDAL BLOCK (Active Comparator): Sonosite machine (M-Turbo) equipped with a large bandwidth, a multifrequency linear probe (6-19 MHz) and needle of diameter and length respectively between 22G and 25G, 35mm and 40mm according to the child's size (Braun).The patient is positioned laterally with their hips flexed to 90°. The sacral hiatus is forming with the two posterior superior iliac spines an equilateral triangle. The puncture is performed between the two sacral cornuae. The sacrococcygeal ligament gives a perceptible 'pop' when crossed. After crossing the sacro-coccygeal ligament, the needle is redirected 30° to the skin surface, and then advanced a few millimeters into sacral canal. After verifying absence of spontaneous reflux of blood or cerebrospinal fluid, slowly injection of Ropivacaine 0.25% 1ml/ kg
  Interventions: Procedure: caudal block
- anterior Quadratus lumborum block (Experimental): Sonosite machine (M-Turbo) equipped with a large bandwidth, a multifrequency linear probe (6-19 MHz) and a 22G, 50-mm, insulated facet type needle (BBraun Stimuplex Ultra 360°). Patients were placed in the lateral position, a probe was placed transversely to the abdominal flank. The needle was inserted using an in-plane technique and was preceded further into the fascia between the QLM and PM. Following confirmation of the correct space with the administration of 0.5-1 ml local anesthetic, block was induced with 1 ml/kg, 0.25% Ropivacaine,
  Interventions: Procedure: anterior Quadratus lumborum block

INTERVENTIONS:
Procedure: anterior Quadratus lumborum block — ultrasound anterior quadratum lumborum block with 1 ml/kg 0.2% ropivacaine
  Arms: anterior Quadratus lumborum block
Procedure: caudal block — ultrasound guided caudal block with 1 ml/kg 0.2% ropivacaine
  Arms: CAUDAL BLOCK

SUMMARY:
Caudal blockade (CB) is one of the most frequently performed regional anaesthetic techniques in children. It's an efficient way to offer perioperative analgesia for painful sub-umbilical interventions but with high incidence of motor block and urinary retention. In one study, psoas compartment block was associated with less morphine comsumption and prolonged duration of analgesia compared to single-shot caudal Block in small children undergoing open hip reduction/osteotomies. Ultasound guided anterior Quadratus lumborum block (AQLB) provides unilateral analgesia to the nerves between the psoas muscle (PM) and the quadratus lumborum muscle (QLM). The first pediatric study evaluating Quadratus lumborum block is encouraging .

The first pediatric study evaluating Quadratus lumborum block is encouraging. To the best of the investigator's knowledge, there are no previously published data comparing the AQLB with other regional techniques in infants undergoing hip surgery.

DETAILED DESCRIPTION:
The aim of this prospective randomized study was to compare the analgesic effects between AQLB and CB in children undergoing unilateral open hip reduction/osteotomies for hip dislocation.

Patients were randomly assigned, into 1 of 2 groups, namely, group CB (n = 20) and group AQLB (n = 20).

Preoperatively all children were premedicated by using oral midazolam (0 .5mg/kg).

anesthesia was induced with 3 to 4% sevoflurane and 50% with 60% nitrous oxide in oxygen.Then fentanyl 3 μg/kg and Propofol 1 - 2mg/Kg were administered for anesthesia induction. Airway was secured with endotracheal tube placed in the mouth facilited by 0.15 mg/kg cistracurium. Anesthesia maintenance was performed with sevoflurane 2% in 50% nitrous oxide.

AQLB and CB were done with 1 ml/kg, 0.25% Ropivacaine (maximum dose limited to 20 ml)

Postoperative follow-up:

All patients received 15 mg/kg paracetamol before extubation. Tramadol 2 mg/kg intravenous was planned as rescue analgesia when CHEOPS score was more than 3. Supplemental IV tramado, 1 mg/kg could be added if necessary every 6 hours.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 2 to 7 years old
* Weight ≤ 20 Kg
* American Society of Anesthesiologists (ASA) physical status I or II
* Planned to undergo unilateral open hip reduction/osteotomies

Exclusion Criteria:

* Cerebral palsy with severe intellectual disability
* Coagulation disorders
* Local or general infection
* Allergy to amide local anesthetics.
* Progressive neurological disorders
* Parenteral refusal
* Spinal dysraphism
* Cutaneous anomalies (angioma, hair truft, naevus or a dimple)near to the puncture

Ages: 2 Years to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2020-03-31 (Actual); Primary Completion 2021-03-30 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
analgesics consumption | day one
  total tramadol consumption

SECONDARY OUTCOMES:
postoperative pain score | day one
  Children's Hospital Eastern Ontario Pain Scale (CHEOPS) [4=no pain ; 13=worst pain]
analgesic rescue | Day one
  time to first analgesic rescue

CONTACTS AND LOCATIONS:
Overall Officials: khaireddine Raddaoui, MD, Principal Investigator — Tunis El Manar University
Locations (1):
- Institut Kassab D'Orthopedie, Tunis, Tunisia